CLINICAL TRIAL: NCT05891288
Title: Sealing of Initial Occlusal Caries in Fissures of Permanent Molars Using Bioactive Versus Fluoride Releasing Fissure Sealants: A Randomized Controlled Trial
Brief Title: Sealing of Initial Occlusal Caries Using Fissure Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer, Department of Conservative Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bioactive fissue sealant
Record Dates: First submitted 2023-05-22; First posted 2023-06-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Caries; Initial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioactive group (Experimental): Bioactive Pits & fissures sealant BioCoat® by Premier®.
  Interventions: Other: BioCoat® by Premier®
- Comparator group (Active Comparator): Fluoride releasing resin based Pits & fissures sealant 3M™ Clinpro™ Sealant
  Interventions: Other: 3M™ Clinpro™ Sealant.

INTERVENTIONS:
Other: BioCoat® by Premier® — Bioactive pits and fissure sealant
  Arms: bioactive group
Other: 3M™ Clinpro™ Sealant. — Fluoride releasing pits and fissure sealant
  Arms: Comparator group

SUMMARY:
The purpose of this study is to compare the performance of newly introduced bioactive resin based pits and fissure sealant versus fluoride releasing resin based pits and fissure sealant in initial carious lesions of fissures in posterior molars in patients at risk of caries. Visual tactile examination and VistaCAM will be used for evaluation.

DETAILED DESCRIPTION:
SmartCap™ Technology, which is used in the novel bioactive fissure sealant, is based on proprietary semi-permeable resin microcapsules. The rechargeable SmartCap microcapsules in BioCoat are packed with ionic fluoride, calcium, and phosphate solutions that diffuse in and out of the sealant. It is hypothesized that fluoride uptake is increased in the presence of calcium and phosphate ions.

With little evidence-based information in the literature about using bioactive fissure sealants to seal initial carious lesions, it was determined that a randomized controlled trial would be beneficial in testing the null hypothesis that bioactive resin pits and fissure sealant will have the same clinical performance as fluoride releasing resin-based pits and fissure sealant in fissures with initial caries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral initial carious fissures in molars showing no signs of caries.
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Sound fissures.
* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Rampant caries.
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of severe bruxism, clenching, or tempromandibular joint disorders.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Retention of sealant | 2 years
  rate of sealant loss

SECONDARY OUTCOMES:
Caries incidence | 2 years
  Rate of caries progression

CONTACTS AND LOCATIONS:
Overall Officials: Omar Shaalan, Principal Investigator — Lecturer, Department of Conservative Dentistry
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelsalam AF, Shaalan O. 24-month efficacy of bioactive versus fluoride sealant for non-cavitated occlusal caries in adults: a randomized clinical trial. Sci Rep. 2025 Dec 11;15(1):43738. doi: 10.1038/s41598-025-29730-8. PMID 41381619